CLINICAL TRIAL: NCT06699355
Title: A Clinical Study to Evaluate the Effect of MK-0616 and Atorvastatin on Their Respective Pharmacokinetics in Healthy Adult Participants
Brief Title: A Study to Evaluate the Drug-Drug Interaction Between Enlicitide Decanoate (MK-0616) and Atorvastatin in Healthy Adult Participants (MK-0616-024)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0616-024; MK-0616-024 (Other: MSD)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atorvastatin (Experimental): Participants receive a single oral dose of atorvastatin (Treatment A) on Day 1.
  Interventions: Drug: Atorvastatin
- Enlicitide Decanoate + Atorvastatin (Experimental): Participants receive a single oral dose of enlicitide decanoate plus a single oral dose of atorvastatin (Treatment B) on Day 1.
  Interventions: Drug: Enlicitide Decanoate; Drug: Atorvastatin
- Enlicitide Decanoate (Experimental): Participants receive a single oral dose of enlicitide decanoate (Treatment C) on Day 1.
  Interventions: Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Enlicitide Decanoate — Oral administration
  Arms: Enlicitide Decanoate; Enlicitide Decanoate + Atorvastatin
Drug: Atorvastatin — Oral administration
  Other Names: Lipitor
  Arms: Atorvastatin; Enlicitide Decanoate + Atorvastatin

SUMMARY:
The goal of this study is to learn what happens to enlicitide decanoate and atorvastatin in a healthy person's body over time. Researchers want to learn what happens to enlicitide decanoate in the body when it is given with and without another medicine called atorvastatin and what happens to atorvastatin in the body when it is given with or without enlicitide decanoate.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, standard and orthostatic vital signs, and electrocardiograms (ECGs)

Exclusion Criteria:

* History of gastrointestinal disease which may affect food and drug absorption or has had a gastric bypass or similar surgery
* History of cancer (malignancy)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Atorvastatin and its Metabolites | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the AUC0-Inf of atorvastatin and its metabolites.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Atorvastatin and its Metabolites | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the AUC0-Last of atorvastatin and its metabolites.
Maximum Plasma Concentration (Cmax) of Atorvastatin and its Metabolites | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Cmax of atorvastatin and its metabolites.
Time to Maximum Plasma Concentration (Tmax) of Atorvastatin and its Metabolites | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Tmax of atorvastatin and its metabolites.
Apparent Terminal Half-Life (t1/2) of Atorvastatin and its Metabolites | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the t1/2 of atorvastatin and its metabolites.
Apparent Clearance (CL/F) of Atorvastatin | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the CL/F of atorvastatin.
Apparent Volume of Distribution (Vz/F) of Atorvastatin | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Vz/F of atorvastatin.
Area Under the Concentration-Time Curve from Time 0 to 24 Hours (AUC0-24hrs) of Enlicitide Decanoate | At designated timepoints (up to approximately 24 hours)
  Blood samples will be collected to determine the AUC0-24hrs of enlicitide decanoate.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the AUC0-Inf of enlicitide decanoate.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the AUC0-Last of enlicitide decanoate.
Maximum Plasma Concentration (Cmax) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Cmax of enlicitide decanoate.
Time to Maximum Plasma Concentration (Tmax) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Tmax of enlicitide decanoate.
Apparent Terminal Half-Life (t1/2) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the t1/2 of enlicitide decanoate.
Apparent Clearance (CL/F) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the CL/F of enlicitide decanoate.
Apparent Volume of Distribution (Vz/F) of Enlicitide Decanoate | At designated timepoints (up to approximately 8 days)
  Blood samples will be collected to determine the Vz/F of enlicitide decanoate.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 10 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com